CLINICAL TRIAL: NCT00357266
Title: Analysis of Differential Gene Expression Profiles in Patients With Defined Ocular Inflammatory Diseases Using CDNA Microarrays and Proteomics
Brief Title: Differences in Genes and Proteins in Active and Controlled Uveitis
Status: Completed | Type: Observational
Sponsor: National Eye Institute (NEI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 020099; 02-EI-0099
Record Dates: First submitted 2006-07-26; First posted 2006-07-27 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2007-10-24

CONDITIONS: Ocular Inflammatory Disease; Uveitis
Keywords: Uveitis; Interleukin 2; Interleukin 2 Receptor; Microarrays; Genetic Expression; Daclizumab; HAT; Zenapax; Proteins; RNA; Ocular Inflammatory Disease
MeSH Terms: conditions — Uveitis; Diabetes Mellitus, Insulin-Dependent, 10

SUMMARY:
This study will examine blood cells and other tissue samples from people with uveitis (eye inflammation) to try to gain a better understanding of this condition. It will look at 1) the differences in cells when uveitis is active and when it is under control; 2) the genes that control the functions of these cells during different stages of the condition; and 3) the proteins the cells make at these different stages.

Patients 6 years of age or older with an eye inflammation of at least 8 weeks' duration may be eligible for this study. They must currently be enrolled in another NEI protocol for evaluation or treatment of uveitis.

Participants will provide blood and possibly eye tissue samples as follows:

Blood samples: Blood samples will be drawn, probably from an arm vein, during periods when the inflammation is bad and when it is quiet. No more than 60 mL (about 4 tablespoons) will be drawn at any visit, and no more than eight samples will be collected in 1 year.

Tissue samples: For patients who require eye surgery, a sample of tissue or fluid that is removed as a routine part of surgery may be provided to investigators in this study for research purposes.

Samples will be collected during patients' visits scheduled as part of their other protocol. The samples will be labeled with a special code number to preserve the patient's identity.

DETAILED DESCRIPTION:
Ocular inflammatory diseases, including uveitis, cause significant visual loss. Previous non-human investigations have identified several cell types, receptor systems and metabolic intermediates that have led to treatment approaches for human patients. However, information on the human genetic expression of these steps in defined inflammatory disease states is lacking. This non-intervention study proposes to obtain peripheral blood and tissue specimens from patients enrolled in other intramural trials for ocular inflammatory diseases and to apply contemporary cDNA microarray technologies for the analysis of differential gene expression. Test results will not be reported to participants or used for diagnostic or therapeutic purposes.

The study's primary objective is to identify unique gene expression profiles as well as disease relevant genes for patients with ocular inflammatory disease at defined clinical stages using cDNA microarray analysis. This will help provide further insight to understand the pathological mechanisms and potential targets for treatment. Some 3,000-5,000 genes will be examined starting with a selected set associated with interleukin (IL) proteins and their receptors, and with tumor necrosis factors (TNF). Purified peripheral blood mononuclear cells (or whole blood lysates using RNA isolation procedures) will be used to isolate total RNA from these samples. Samples will be taken during periods of active or recurring inflammatory disease and again during periods of quiescence after treatment. The microarray tools and methods for genetic analysis are now available both at NEI and the collaborating NIA laboratories.

A secondary objective is to analyze the circulating protein profiles in serum or other available tissue or fluid specimens from patients with ocular inflammatory disease at the same time points as described above. These samples will be analyzed using 2-dimensional SDS-PAGE for profiling proteomic differences in patients at defined clinical stages. In-gel digestion and subsequent sequence analysis by mass spectroscopy will be performed if differentially expressed protein(s) of interest are to be identified. Other methods such as flow cytometry analysis and proliferation assays using purified PBMCs will be used to examine expression status of cell surface markers of interest (e.g., CD25) as well as responses to antigen and mitogens at the peak and trough serum concentrations of daclizumab therapy.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Participant is 6 or more years of age.
  2. Participant has a diagnosis of an ocular inflammatory disease of at least eight weeks' duration prior to enrollment, requiring medical treatment to control the ocular inflammation. This treatment must require using a corticosteroid (e.g., prednisone or equivalent) or an investigational treatment, or any combination of two or more anti-inflammatory treatments, including for example prednisone, cyclophosphamide, cyclosporine, azathioprine, mycophenolate mofetil, methotrexate, etc. Participants are anticipated to have, but are not restricted to, the following conditions: scleritis, intermediate or posterior uveitis, intermediate uveitis of the pars planitis subtype, sarcoidosis, the Vogt-Koyanagi-Harada (VKH) syndrome, Behcet's disease, juvenile rheumatoid arthritis (JRA), retinal vasculitis or sympathetic ophthalmia.
  3. Participant is currently enrolled in another NEI protocol for one of the above (or related) conditions that requires periodic visits to NIH for treatment and/or evaluation.
  4. Participant is able to understand and sign an informed consent (or applicable assent) and if the participant is younger than the age 18 at enrollment, has a parent or legal guardian who is able to understand and sign a consent form on their behalf.

EXCLUSION CRITERIA:

1. Participant is under the age of 6 years.
2. Participant has inadequate vascular access to obtain a routine venous peripheral whole blood specimen totaling up to 50 mL at a single visit.
3. Participants has an inadequate peripheral leukocyte count such that it would be unlikely to provide an adequate RNA sample. For this purpose, a total leukocyte count below 3 x 10(9)/L will exclude a participant at enrollment. Unless there is a recognized medical condition likely to reduce leukocyte counts, blood counts from a prior visit up to 5 weeks earlier may be used to determine eligibility for a first or subsequent sample collection. (A participant who initially enrolls with an adequate leukocyte count may remain enrolled if counts subsequently fall below the limit, but will not have blood samples drawn for this protocol until the leukocyte count recovers above the limit).

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60
Dates: Start 2002-02-01; Study Completion 2007-10-24

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Schena M, Shalon D, Davis RW, Brown PO. Quantitative monitoring of gene expression patterns with a complementary DNA microarray. Science. 1995 Oct 20;270(5235):467-70. doi: 10.1126/science.270.5235.467. PMID 7569999